CLINICAL TRIAL: NCT00000887
Title: A Phase I Trial of the Safety, Tolerance, and Pharmacokinetics of Oral Nelfinavir (Viracept) Co-Administered With Zidovudine (ZDV) and Lamivudine (3TC) in HIV Infected Pregnant Women and Their Infants
Brief Title: A Study to Evaluate the Safety and Tolerance of Nelfinavir (NFV) Given With Zidovudine (ZDV) and Lamivudine (3TC) in HIV-Positive Pregnant Women and Their Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 353; 10603 (Registry Identifier: DAIDS ES); PACTG 353
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Pregnancy
Keywords: Pregnancy; Pregnancy Complications, Infectious; Drug Therapy, Combination; Zidovudine; HIV Protease Inhibitors; Lamivudine; Disease Transmission, Vertical; Nelfinavir; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious | interventions — Nelfinavir; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Nelfinavir mesylate
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
The purpose of this study is to see if giving nelfinavir (NFV) plus zidovudine (ZDV) plus lamivudine (3TC) to HIV-positive pregnant women and their babies is safe. This study will also look at how long these drugs stay in the blood.

ZDV has been given to mothers in the past to reduce the chances of passing HIV on to their babies. However, better treatments are needed to further reduce these chances and to better suit the treatment needs of mothers and their children. Taking a combination of anti-HIV drugs during pregnancy may be an answer.

DETAILED DESCRIPTION:
Despite the dramatic reduction of perinatal HIV transmission by the administration of ZDV to mother and infant, new and more potent strategies are needed to further reduce perinatal transmission and better suit the diverse treatment needs of these patients. Initiation of triple antiretroviral combinations during gestation, particularly combinations that include drugs that cross the placenta such as 3TC, may be the most effective in reducing maternal virus load to its lowest levels prior to delivery.

Women receive nelfinavir plus 3TC plus ZDV antepartum (Study Day 0 until onset of active labor) through postpartum (after cord clamped to 12 weeks). [AS PER AMENDMENT 10/28/97: If patient presents in active labor with less than 1 hour to delivery time, the institutional protocol for ZDV infusion during labor should be followed.] [AS PER AMENDMENT 1/26/99: For maternal dosing, one Combivir tablet bid can be substituted for the individual formulation of 3TC and ZDV. For mothers who receive Combivir during the antepartum period, Combivir is held during labor and delivery, and the separate formulations of ZDV and 3TC are used. Patients who prematurely discontinue study treatment should continue to be followed on study for the duration of the study.] Full pharmacokinetic sampling is performed 10 to 15 days after start of therapy [AS PER AMENDMENT 2/7/00: 10 to 15 days after study entry for women currently taking nelfinavir] and again 5 to 6 weeks after delivery. A maternal blood sample and cord blood sample is collected at birth for analysis of nelfinavir concentrations. Maternal HIV RNA in plasma is monitored throughout the study. Cervicovaginal secretions are collected at entry, late gestation, and postpartum to assess the presence of HIV. A single pharmacokinetics sample is collected with each cervicovaginal secretion. Serial CD4/CD8 activation markers are measured in women during gestation and postpartum. Infants receive nelfinavir plus 3TC plus ZDV beginning approximately 12 hours following birth and continuing for 6 weeks. After birth, several blood samples are collected from the infant for determination of washout kinetics of nelfinavir. Full pharmacokinetics sampling is performed 5 to 8 days post birth and 5 to 6 weeks following multiple doses. Pharmacokinetic samples are analyzed on the first six mother-infant pairs and dosing may be adjusted accordingly for the next cohort. Agouron has agreed to make nelfinavir available to all interested study participants for a period of 6 months after the study via the patient assistance program.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are at least 13 years old (need consent of parent or guardian if under 18).
* Are HIV-positive.
* Are in the 2nd or 3rd trimester (14 to 34 weeks pregnant) and are pregnant with one or two children.
* Have a normal ultrasound exam.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Cannot take ZDV or 3TC.
* Have an active opportunistic (HIV-associated) or bacterial infection, or a severe medical condition.
* Have severe diarrhea.
* Are at risk for premature birth or pregnancy complications.
* Have a family history of phenylketonuria (PKU).
* Plan to breast-feed.
* Abuse alcohol or drugs.
* Cannot visit the same clinic for the duration of the study.
* Have taken certain anti-HIV drugs.

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24
Dates: Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Bryson, Study Chair; Mark Mirochnick, Study Chair; Alice Stek, Study Chair
Locations (7):
- United States (7):
  - Usc La Nichd Crs, Los Angeles, California
  - Tulane Univ. Health Science Ctr., Tulane Univ. Hosp. & Clinic, New Orleans, Louisiana
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Johns Hopkins Hosp. & Health System - Dept. of Peds., Div. of Infectious Diseases, Baltimore, Maryland
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - UNC at Chapel Hill School of Medicine - Dept. of Peds., Div. of Immunology & Infectious Diseases, Chapel Hill, North Carolina
  - St. Christopher's Hosp. for Children, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Bryson Y, Stek A, Mirochnick M, et al. Pharmacokinetics, antiviral activity, and safety of nelfinavir (NFV) with ZDV/3TC in pregnant HIV-infected women and their infants. PACTG 353 cohort 2. 9th Conference on Retroviruses and Opportunistic Infections. 2002, February 24-28; Seattle Washington (abstract no 795)
- [Result] Bryson YJ, Mirochnick M, Stek A, Mofenson LM, Connor J, Capparelli E, Watts DH, Huang S, Hughes MD, Kaiser K, Purdue L, Asfaw Y, Keller M, Smith E; PACTG 353 Team. Pharmacokinetics and safety of nelfinavir when used in combination with zidovudine and lamivudine in HIV-infected pregnant women: Pediatric AIDS Clinical Trials Group (PACTG) Protocol 353. HIV Clin Trials. 2008 Mar-Apr;9(2):115-25. doi: 10.1310/hct0902-115. PMID 18474496